CLINICAL TRIAL: NCT00098085
Title: A Phase II Study of the Feasibility to Derive Autologous Vaccine (HSPPC-96) From Tumor Tissue for Clinical Administration in Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: Study of the Feasibility to Derive Vaccine From Tumor Tissue in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: C-100-26
Record Dates: First submitted 2004-12-03; First posted 2004-12-06 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Non-Small-Cell Lung Carcinoma; Lung Cancer; Pulmonary Cancer
Keywords: Lung cancer; Non-small cell lung cancer; Pulmonary; Immunotherapy; Vaccine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — vitespin

INTERVENTIONS:
Biological: HSPPC-96

SUMMARY:
Antigenics is enrolling patients in a Phase II study testing the feasibility to derive an autologous investigational vaccine (HSPPC-96) from the tumor tissue of patients with resectable non-small cell lung cancer.

Vaccine production will be attempted on all patients who undergo surgery and meet all inclusion/exclusion criteria.

DETAILED DESCRIPTION:
Antigenics is enrolling patients in a Phase II study testing the feasibility to derive an autologous investigational vaccine (HSPPC-96) from the tumor tissue of patients with resectable non-small cell lung cancer.

All patients will undergo surgery to remove the tumor and will be followed for recurrence and overall survival.

The primary goal of this trial is to determine if HSPPC-96 can be made from the tumor tissue of patients with resectable non-small cell lung cancer.

The secondary goals are to further characterize the safety and efficacy profile, to evaluate disease recurrence in patients receiving, and to evaluate overall survival in patients receiving HSPPC-96.

HSPPC-96 is an investigational, immunotherapeutic agent made from an individual patient's own tumor, which is collected at the time of surgery. A portion of the tumor tissue is sent to Antigenics' manufacturing facility where it will undergo processing to create a vaccine. This vaccine may help the patient's immune system attack cancerous cells while leaving healthy cells alone.

ELIGIBILITY:
This is a summary of criteria. Only the Principal Investigator can determine eligibility.

Inclusion Criteria:

* Suspected non-small cell lung cancer, Stage IB, Stage II, or Stage IIIA
* Tumor size > 3x3 cm or equivalent to a 9 cm² lesion
* Scheduled surgery with curative intent
* At least 18 years of age
* Must not be pregnant or breast feeding
* Agree to not receive any other investigative agent at any time while enrolled in this study

Exclusion Criteria:

* Previous treatment for non-small cell lung cancer
* Clinical signs or symptoms of brain metastases
* History of immune suppression or autoimmune disorder
* Severe active infection or other serious medical illness, that in the opinion of the Principal Investigator, would prevent study completion
* Other malignancies in the past 5 years, except adequately treated in situ cervix carcinoma or non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-09; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary goal of this trial is to determine if HSPPC-96 can be made from the tumor tissue of patients with resectable non-small cell lung cancer.

SECONDARY OUTCOMES:
The secondary goals are to further characterize the safety and efficacy profile, to evaluate disease recurrence in patients, and to evaluate overall survival in patients receiving HSPPC-96.

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom